CLINICAL TRIAL: NCT05066243
Title: Development and Psychometric Analysis of a Patient Reported Outcome Measure for Patients Attending a Specialist Vulval Clinic
Brief Title: A Patient Reported Outcome Measure for Vulval Conditions
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Liverpool University Hospitals NHS Foundation Trust (Other Government)
Responsible Party: Sponsor
Other Study IDs: 6059
Record Dates: First submitted 2021-09-23; First posted 2021-10-04 (Actual); Last update posted 2021-10-04 (Actual); Status verified 2020-10

CONDITIONS: Vulval Dermatoses; Vulval Pain Syndromes
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- focus group: 15 service users for focus group
- questionnaire: 150 patients to test questionnaire
  Interventions: Other: questionnaire

INTERVENTIONS:
Other: questionnaire — this study is to develop a questionnaire for vulval conditions
  Groups: questionnaire

SUMMARY:
To create a new patient reported outcome measure in the form of a questionnaire, which will accurately reflect the profound impact that vulval dermatoses and vulval pain syndromes have on patients' quality of life

DETAILED DESCRIPTION:
In order to create the proposed vulval specific patient reported outcome measure we will use semi structured questionnaires and a focus group interview.

Methods:

Participating patients will be recruited through their attendance at a specialist vulval dermatology clinic across two secondary care centres, by the direct patient care team. Written consent will be obtained at every stage and each patient will receive written information in the form of a patient information leaflet as to why the research is being conducted. Patients will be reassured that declining involvement in the research will have no impact upon the quality of their care and that their involvement is entirely voluntary.

Initially fifty (50) follow up/new patients attending the specialist vulval clinic across two sites will be invited to answer questionnaires on their attendance at clinic, which will ask a number of open-ended questions about aspects of their vulval condition that may have affected them. These questions have been devised by the research team based on professional experience and the results of previous research, which have identified common themes to life impairment to include symptoms, sexual function, personal relationships, emotions, daily activities and social/leisure activities.4,7 Based upon the findings we will develop a preliminary questionnaire (patient reported outcome measure) in conjunction with an expert panel compromising of a consultant dermatologist and speciality doctor in gynaecology, both of which have a specialist interest in vulval medicine. This questionnaire will be subsequently piloted on a focus group of fifteen (15) patients with a variety of vulval conditions. The research team feels that a small focus group would be preferential over individual interviews as we hope a group discussion in which people can share their experiences will stimulate discussion, generate new ideas and help reach a consensus opinion on the newly created patient reported outcome measure. Furthermore, focus groups have been successfully used in other studies of patients suffering with vulval disease. 8,9 Individual diagnoses will not be discussed in the patient group setting and It will be attended by the full patient care team and directed by the Chief Investigator. Based upon their comments and professional consensus the questionnaire will be further refined. Patients will be consented for their involvement and the justification of the research explained. These patients may or may not have been asked to complete the original questionnaire which was used to help develop the subsequent patient reported outcome measure.

In order to authenticate the newly created patient outcome measure, one hundred (100) patients attending the specialist vulval dermatology clinic on an opportunistic basis across two centres (both new and follow up) will be invited to participate in completing the newly created questionnaire. These patients may be previously been part of the pilot group and/or been asked to contribute to the initial questionnaire which led to the development of the patient reported outcome measure. All patients will be given the questionnaire fifteen (15) minutes prior to their clinic appointment and given the opportunity to ask questions in their clinic appointment should they wish.

A second duplicate questionnaire will be given to all the participating women in a self-addressed envelope, with instructions to complete it after two weeks and return it in the post. If the second questionnaire is not received within three weeks, two reminder calls will be made. Through repeating the questionnaire at 2 weeks, its reliability can be determined using statistical methods.

At the same clinic visit patients will also be asked to complete the dermatology life quality index (DLQI), which is a questionnaire that is routinely used in clinical practice to assess the impact of a patient's skin condition on their quality of life. This is done so comparisons can be made between the DLQI and new questionnaire. Statistical methods will be used analyse the results and interpret the authenticity of the new questionnaire.

Data analysis

The validation of the vulval specific patient reported outcome measure will be addressed in a number of ways:

The test retest reliability will be assessed by asking the women to fill out the same questionnaire two weeks after their initial recruitment into the study. The second questionnaire will be given to the women with a self-addressed envelope after their initial recruitment into the study, with instructions to complete it after two weeks and return it in the post. This time period was chosen in order to avoid recall bias. If a second questionnaire is not received in three weeks, two reminder calls will be places. Test-retest reliability will be measured for individual questions using the kappa coefficient for individual questions. The test retest reliability for the sum of the different scales will be measured by intra class coefficients. Cronbach's alpha will be used to measure internal consistency.

Confirmatory factor analysis will be used to verify the five a priori scales of the vulval specific patient reported outcome measure. (These are assumed to be sexual function, emotions, symptoms, daily activities and social functioning) This will be used to address construct validity.

Construct validity will be also be determined through testing against the Dermatology Quality Life Index. There is currently no gold standard quality of life measure used in vulval conditions, but the DLQI is used routinely in dermatology practice, including patients who present to the specialist vulval clinic. All patients (n=100) will be given a DLQI form to complete at the same time as the piloted questionnaire.

ELIGIBILITY:
Inclusion Criteria:

* 1) Adult female patients aged 18 upwards 2) Patients must have a vulval dermatosis or vulval pain syndrome confirmed on history and examination. These will include inflammatory dermatoses, non-inflammatory dermatoses and vulval pain syndromes

Exclusion Criteria:

* 1) Patient with a vulval condition thought to be of a sexually transmitted aetiology 2) Patients lacking capacity

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: vulval dermatoses and vulval pain syndromes patients
Sampling Method: Non-Probability Sample
Enrollment: 165 (Estimated)
Dates: Start 2021-10-09 (Estimated); Primary Completion 2022-02-01 (Estimated); Study Completion 2022-04-15 (Estimated)

PRIMARY OUTCOMES:
questionnaire development | 1 year
  questionnaire development

IPD SHARING:
Plan to Share IPD: Undecided